CLINICAL TRIAL: NCT05979051
Title: A Multicenter, Single-arm/Randomized, Double-blind, Active-controlled, Parallel-group Phase 2/3 Clinical Study to Evaluate the Efficacy and Safety of SHR-1703 for Patients With EGPA
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR-1703 in Subjects With Eosinophilic Granulomatosis With Polyangiitis （EGPA）
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHR-1703-301
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: A single-arm/randomized, double-blind, placebo-controlled, parallel-group Phase 2/3 clinical study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR-1703
  Interventions: Drug: SHR-1703
- Mepolizumab Injection (Active Comparator): SHR-1703 Placebo
  Interventions: Drug: Mepolizumab Injection

INTERVENTIONS:
Drug: SHR-1703 — SHR-1703 will be administered by Subcutaneous injection in Phase 2 and Phase 3.
  Arms: Treatment group A
Drug: Mepolizumab Injection — Mepolizumab Injection and Matching Placebo will be administered by Subcutaneous injection in Phase 3
  Arms: Mepolizumab Injection

SUMMARY:
This study is a phase 2/3 clinical trial to evaluate the efficacy and safety of SHR-1703 in patients with EGPA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 18 years or older;
2. Diagnosed with EGPA for at least 6 months;
3. History of relapsing or refractory EGPA；
4. Stable dose of oral prednisone of ≥7.5 mg/day (but not >50 mg/day) for at least 4 weeks prior to randomization;
5. If receiving immunosuppressive therapy (excluding cyclophosphamide), the dosage must be stable within 4 weeks prior to randomization and during the study.

Exclusion Criteria:

1. Subjects with other eosinophilic-related diseases;
2. Diagnosed with granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA).
3. Life-threatening EGPA within 3 months prior to randomization;
4. Malignancy history within 5 years prior to randomization;
5. Immunodeficiency;
6. Uncontrolled hypertension；
7. Uncontrolled cerebrovascular and cardiovascular disease;
8. parasitic infection within 6 months prior to randomization;
9. Active infectious disease requiring clinical treatment within 4 weeks prior to randomization;
10. Subjects with a dose of oral prednisone of >50 mg/day within 4 weeks prior to randomization;
11. Oral or intravenous cyclophosphamide therapy within 4 weeks prior to randomization;
12. Intravenous or subcutaneous immunoglobulin within 12 weeks prior to randomization;
13. Biological agents or TH2 cytokine inhibitors used within 12 weeks prior to randomization or within 5 half-lives of the drug;
14. Rituximab used within 6 months prior to randomization；
15. Surgical plans that might affect the evaluation;
16. Significant laboratory abnormalities；
17. Prolonged QTc interval or other electrocardiogram abnormalities with significant safety risk at screening;
18. History of drug or substance abuse or alcohol abuse within 1 year prior to screening;
19. Subjects participated another clinical study and received active drug within 30 days or 5 half-lives of the drug prior to screening;
20. Subjects is pregnant, lactating, or planning to be pregnant;
21. Subjects have a known history of hypersensitivity or intolerance to anti-IL-5 mabs or other biological agents or previous failure of IL-5/IL-5R therapy;
22. Other conditions unsuitable for participation in the study per investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in oral glucocorticoid dose (OCS) | Up to week 12
  Phase 2
The Proportion of subjects in EGPA remission | week 36 and week 48
  Phase 3

SECONDARY OUTCOMES:
Change from baseline in oral glucocorticoid dose | Up to week 24, week 48
  Effectiveness Indicators (Phase 2)
The proportion of subjects with OCS dosage ≤5 mg/d | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The proportion of subjects with at least 50% reduction of OCS dosage from baseline | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The Proportion of subjects with EULAR remission | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The Proportion of subjects achieving EULAR remission at week 12 and week 24 of treatment and maintaining it up to week 48 | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The Proportion of subjects with EGPA remission | week 24, week 48
  Effectiveness Indicators (Phase 2)
The proportion of subjects achieving EGPA remission within 24 weeks of treatment and maintaining it up to week 48 | week 24, week 48
  Effectiveness Indicators (Phase 2)
The proportion of subjects with EGPA relapse | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The time to the first relapse of EGPA | Up to week 48
  Effectiveness Indicators (Phase 2)
The proportion of subjects with Severe relapse of EGPA | week 12, week 24, week 48
  Effectiveness Indicators (Phase 2)
The time of the first Severe relapse of EGPA | Up to week 48
  Effectiveness Indicators (Phase 2)
Changes from baseline in Pre- and post-Bronchodilator FEV1 | Up to week 48
  Effectiveness Indicators (Phase 2)
The Proportion of subjects with EULAR remission | week 36, week 48
  Effectiveness Indicators (Phase 3)
The Proportion of subjects with EGPA remission | week 36, week 48
  Effectiveness Indicators (Phase 3)
The Proportion of subjects achieving EULAR remission within 24 weeks of treatment and maintaining it up to week 48 | week 24, week 48
  Effectiveness Indicators (Phase 3)
The proportion of subjects achieving EGPA remission within 24 weeks of treatment and maintaining it up to week 48 | week 24, week 48
  Effectiveness Indicators (Phase 3)
Cumulative weeks of EGPA remission through week 48, categorized as 0 weeks; >0 to <12 weeks; 12 to <24 weeks; 24 to <36 weeks; or ≥36 weeks | week 0, week 12, week 24, week 36, week 48
  Effectiveness Indicators (Phase 3)
Change from baseline in OCS | Week 24, Week 48
  Effectiveness indicators (Phase 3)
The proportion of subjects with OCS dosage ≤5 mg/d | week 24, week 48
  Effectiveness indicators (Phase 3)
The proportion of subjects with at least 50% reduction of OCS dosage from baseline | week 24, week 48
  Effectiveness indicators (Phase 3)
The Proportion of subjects with EGPA relapse | week 24, week 48
  Effectiveness indicators (Phase 3)
The Proportion of subjects with Severe relapse of EGPA | week 24, week 48
  Effectiveness indicators (Phase 3)
The time to the first relapse of EGPA | Up to week 48
  Effectiveness indicators (Phase 3)
The time of the first Severe relapse occurred of EGPA | Up to week 48
  Effectiveness indicators (Phase 3)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided